CLINICAL TRIAL: NCT04181541
Title: Can Midlevel Providers Manage Medical Abortion in the Second Trimester as Safely and Effectively as Physicians? A Randomized Controlled Trial in Ethiopia
Brief Title: Midlevel Versus Physician-provided Medical Abortion in the Second Trimester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ipas (Other)
Collaborators: St. Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM23/146
Record Dates: First submitted 2019-11-22; First posted 2019-11-29 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Induced Abortion; Second Trimester Abortion; Medical Abortion; Health Personnel
Keywords: Midlevel provider

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized, controlled, non-inferiority study comparing management of medical abortion by either nurse midwives or physicians for women undergoing induced abortion at a gestational ages > 13 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women receiving abortion care by physicians (Active Comparator): Patients who receive second trimester medical abortion care from a physician.
  Interventions: Procedure: Provider type: Physicians
- Women receiving abortion care from midlevel providers (Experimental): Patients who receive second trimester medical abortion care from a midlevel provider.
  Interventions: Procedure: Provider type: Midlevel Providers

INTERVENTIONS:
Procedure: Provider type: Physicians — In this cohort, women will receive second trimester medical abortion care from physicians
  Arms: Women receiving abortion care by physicians
Procedure: Provider type: Midlevel Providers — In this cohort, women will receive second trimester medical abortion care from midlevel providers.
  Arms: Women receiving abortion care from midlevel providers

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of second trimester medical abortion when provided by nurse midwives compared with physicians. The study sample will be obtained from Michu Clinic, affiliated with St Paul's hospital, in Addis Ababa.

DETAILED DESCRIPTION:
About 10% of all abortions globally take place at or after 13 weeks gestation. Women seeking second-trimester abortion services are often the most vulnerable and socially disadvantaged population.Studies show the rate of second-trimester abortion procedures remains stable over time, even in high-access locations, confirming the ongoing need for accessibility to services in rural locations with limited access to care. In Ethiopia, second-trimester abortion services are widely available in Addis Ababa, making up a high proportion of the total number of abortions occurring each year in the country; however, access to accurate and reliable data is limited.

The World Health Organization recommends that abortion can be provided at the lowest level of the healthcare system (WHO abortion guidelines). Training mid-level providers, such as midwives, nurses and other non-physician providers, to conduct second trimester aspiration abortions is proposed as a way to increase women's access to safe abortion procedures and has been highlighted by the WHO as an area in which rigorous research is needed (WHO task-sharing guidelines).

The investigators seek to conduct a comparative study of patients undergoing second trimester medical abortion provided by either physicians or nurse midwives.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give consent for participation
* Intrauterine pregnancy with confirmed gestational age >13 weeks and <20 weeks
* Presenting for induced abortion at Michu Clinic
* Speaker of Amharic or Oromo

Exclusion Criteria:

* Women unable to give consent for participation
* Gestational age <13 or >20 weeks
* Adolescents aged less than 16 years
* Women with an allergy to or contraindications to mifepristone or misoprostol
* Women with a history of more than one previous hysterotomy
* Women seeking treatment for incomplete abortion, intrauterine fetal demise, or postabortion care
* Women with chronic hypertension or adrenal failure
* Women on chronic steroid treatment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Time to expulsion | Time (hours/minutes) from first dose of misoprostol until the fetus is expelled, up to 72 hours
  Time to expulsion of fetus after medical abortion regimen initiated

SECONDARY OUTCOMES:
Total number of misoprostol doses | Time (hours/minutes) from first dose of misoprostol until the fetus and placenta are expelled, up to 72 hours
  Doses of misoprostol needed for completion of abortion
Need for ultrasound to confirm gestational age | At the time of eligibility for the abortion is assessed, need for confirmatory ultrasound recorded (up to 1 day)
  Whether ultrasound was needed to estimate gestational age
Need for intervention by a physician | Assessed at the time of discharge and reflecting entire duration of hospitalization (up to 7 days)
  whether any physician involvement was needed to manage the case (from nurse-led services)
Serious complications/ morbidity | Assessed at the time of discharge and reflecting entire duration of hospitalization (up to 7 days)
  Whether the following complications occur while a patient is receiving abortion services: hemorrhage requiring transfusion, placental retention requiring removal, uterine rupture, fever/ signs of infection requiring antibiotic treatment.
Adverse events | up to 7 days after discharge
  Whether adverse events occurred that required a return to the hospital after discharge from Michu clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Kapp, MD, MPH, Principal Investigator — Ipas
Locations (1):
- St. Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No